CLINICAL TRIAL: NCT04488198
Title: Acupuncture in Pediatrics and Adolescents With Chronic Inflammatory Bowel Diseases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christina Hafner, Christina Hafner, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1773/2018
Record Dates: First submitted 2020-06-26; First posted 2020-07-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Morbus Crohn; Colitis, Ulcerative
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): 20 CIBD patients do not receive acupuncture or placebo-acupuncture.
- Acupuncture group (Active Comparator): 20 CIBD patients receive 8 sessions of acupuncture therapy with 0,3 x 30mm needles (asia-med special number 16).
  Interventions: Other: Acupuncture
- Placebo group (Placebo Comparator): 20 CIBD patients receive 8 sessions of sham acupuncture with placebo-needles 0,3 x 30mm (Streitberger).
  Interventions: Other: Placebo-Acupuncture

INTERVENTIONS:
Other: Acupuncture — Patients receive 8 acupuncture sessions (1 session per week, 20 minutes per session) with acupuncture needles.
  Arms: Acupuncture group
Other: Placebo-Acupuncture — Patients receive 8 acupuncture sessions (1 session per week, 20 minutes per session) with placebo-needles.
  Arms: Placebo group

SUMMARY:
Chronic inflammatory bowel disease (CIBD) with its prevalence of 2.6 million people in Europe is diagnosed in 25% before the age of 18 years. Early remission is intended to improve child growth, quality of life and reduce psychological comorbidities. Additionally to conventional drugs one third of pediatric CIBD patients use alternative treatment strategies. However, there is a lack of evidence of acupuncture as complementary medicine in pediatric CIBD on the disease activity and inflammation. Therefore, the main aim of this study is to evaluate the effect of acupuncture in children with CIBD on the Pediatric Ulcerative Colitis Activity Index (PUCAI) and the Weighted Pediatric Crohn's Disease Activity Index (sPCDAI), which are non-invasive validated instruments to measure the disease activity. Furthermore, this study aims to investigate the effect of acupuncture on chronic pain, quality of life and parameters of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* mild/moderate CIBD
* stable pharmacological treatment at least for 8 weeks

Exclusion Criteria:

* complementary alternative medicine

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Activity Index | At beginning vs 8 weeks
  Disease Activity Index (either Paediatric Ulcerative Colitis Activity Index in case of patients with ulcerative colitis or Weighted Pediatric Crohn's Disease Activity in patients with Crohn's disease)
Disease Activity Index | At beginning vs 4 weeks
  Disease Activity Index (either Paediatric Ulcerative Colitis Activity Index in case of patients with ulcerative colitis or Weighted Pediatric Crohn's Disease Activity in patients with Crohn's disease)

SECONDARY OUTCOMES:
Quality of Life in Children and Adolescents measured by KINDL(R) | At beginning vs 4 weeks
  The quality of life will be measured using the KINDL(R) questionnaire. The data will be transformed according to the manual of the questionnaire. The total score of quality of life ranges from 0 to 100. A higher score is associated with a better quality of life.
Quality of Life in Children and Adolescents measured by KINDL(R) | At beginning vs 8 weeks
  The quality of life will be measured using the KINDL(R) questionnaire. The data will be transformed according to the manual of the questionnaire. The total score of quality of life ranges from 0 to 100. A higher score is associated with a better quality of life.
Quality of Life in Children and Adolescents measured by ILK | At beginning vs 4 weeks
  The quality of life will be also measured using the ILK questionnaire (Inventar zur Erfassung der Lebensqualität bei Kindern und Jugendlichen). The total score of quality ranges from 0 to 28. A higher score is associated with a better quality of life.
Quality of Life in Children and Adolescents measured by ILK | At beginning vs 8 weeks
  The quality of life will be also measured using the ILK questionnaire (Inventar zur Erfassung der Lebensqualität bei Kindern und Jugendlichen). The total score of quality ranges from 0 to 28. A higher score is associated with a better quality of life).
Pain assessment | At beginning vs 4 weeks
  The pain will be measured using the numerating scale, which ranges from 0 (no pain) to 10 (worst pain possible).
Pain assessment | At beginning vs 8 weeks
  The pain will be measured using the numerating scale, which ranges from 0 (no pain) to 10 (worst pain possible).
C reactive protein | At beginning vs 4 weeks
  As one parameter of inflammation the C reactive protein will be measured in mg/dl.
C reactive protein | At beginning vs 8 weeks
  As one parameter of inflammation the C reactive protein will be measured in mg/dl.
Leukocytes | At beginning vs 4 weeks
  As another parameter of inflammation the leukocytes will be measured in 10^9/L
Leukocytes | At beginning vs 8 weeks
  As another parameter of inflammation the leukocytes will be measured in 10^9/L
Erythrocyte sedimentation rate | At beginning vs 4 weeks
  As another inflammatory parameter the erythrocyte sedimentation rate (mm/hour) will be measured.
Erythrocyte sedimentation rate | At beginning vs 8 weeks
  As another inflammatory parameter the erythrocyte sedimentation rate (mm/hour) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Scharbert, MD, Principal Investigator — MedUniVienna
Locations (1):
- Department of Anesthesia, General Intensive Care and Pain Management,Medical University of Vienna, Vienna, Austria